CLINICAL TRIAL: NCT03608410
Title: ProWide - Patient Reported Outcomes Used for Weekly Internet-based DEtection of Progressive Disease in Lung Cancer; a Randomized Controlled Trial
Brief Title: Intensified Follow-up of Lung Cancer Using Weekly Questionnaires Via the Internet
Acronym: ProWide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regional Hospital West Jutland (Other)
Collaborators: Danish Cancer Society (Other); Danish Lung Cancer Group (Other)
Responsible Party: Principal Investigator, Rasmus Blechingberg Friis, MD, Principal Investigator, Regional Hospital West Jutland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ProWide; R184-A11805-17-S57 (Other Grant/Funding Number: Danish Cancer Society); 2017-41-5251 (Registry Identifier: Danish Data Protection Agency)
Record Dates: First submitted 2018-07-11; First posted 2018-08-01 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Lung Cancer
Keywords: Patient reported outcomes; Internet; TelePRO
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: The randomization will be done by the AmbuFlex-system (a generic on-line system for self-recorded patient reported outcomes) as a part of the inclusion process.
  A text message reminder is sent weekly for patients in the intervention group by the system.
  Quality of Life questionnaires will automatically be sent via a safe internet connection to participants in both groups every 2 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRO intervention (Experimental): Weekly PRO questionnaires Quality of life every 2 months
  Interventions: Other: Weekly Internet based PRO questionnaires
- Standard of care (No Intervention): Quality of life every 2 months

INTERVENTIONS:
Other: Weekly Internet based PRO questionnaires — If core symptoms worsen and exceeds a predefined threshold, a PRO-notification is sent to the hospital.
  Arms: PRO intervention

SUMMARY:
This randomized controlled trial (RCT) will test if weekly supplementary internet-based self-monitoring of 12 core symptoms can increase survival in Danish lung cancer patients during follow-up or maintenance treatment. A threshold mechanism will automatically send an alert to the hospital in case of alarming or worsening symptoms and the patient will be contacted by the treating clinicians.

DETAILED DESCRIPTION:
This multicenter RCT study enrolls patients diagnosed with stage IV og incurable stage III lung cancer who has non-progressive disease at first evaluation scan. Patients in follow-up or maintenance therapy are eligible.

492 patients will be included in the study with 246 patients in each group.

Intervention In the experimental arm, patients will be asked to fill in a web-based Patient Reported Outcome (PRO) questionnaire every week. If one of the reported symptoms worsens and exceed a predefined threshold of severity, a notification is automatically sent to the hospital. A nurse will review til questionnaire and contact the patient for verification of symptoms. If progression of disease is suspected, a CT scan will be made. Otherwise, the nurse will schedule a visit at the clinic for physical examination and evaluation by a clinician. If progressive disease is not suspected, supportive care will be adjusted and the patient will continue follow up according to the usual schedule.

The interventions ends in case of progressive disease.

Evaluation Baseline CT-scan of thorax and upper abdomen is performed prior to initial treatment and an evaluation CT scan at the time of enrolment. CT scans will be repeated for assessing signs of progression due to standard follow-up procedures in both groups. If progressive disease is suspected based on symptom development, the following scan will be rescheduled to as soon as possible.

Quality of life (QoL) will be measured in both groups using EORTC (European Organisation for Research and Treatment of Cancer) QOL-C30 / LC13 and HADS (Hospital Anxiety And Depression Scale) quality of life questionnaires every 2 month during the study period.

Objectives The primary objective is to test if supplementary weekly PRO monitoring increases overall survival in a Danish Lung Cancer population

Monitoring Clinical decisions taken on the basis of PRO notifications will daily be registered in the software system by the clinicians. Patient responses to questionnaires and PRO-notification handling by the clinical staff will be monitored by Primary Investigator.

End points will be entered by local site investigators.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with lung cancer (NSCLC and SCLC), who have received 1st line induction treatment* for lung cancer and have no sign of progressive disease at first evaluation CT scan.
2. Patients diagnosed with stage III treated with palliative intention, and stage IV, regardless of treatment intention.
3. Diagnosis proven by cytology or histology
4. Age ≥ 18 years
5. Performance status (PS) ≤ 2 within 15 days before enrolment
6. First evaluation CT scan performed within four weeks from enrolment
7. Patient with acess to internet, Mobile phone and E-boks (Danish digital secure mail system)
8. Patient has given his/her written informed consent before any specific procedure from protocol

   * Induction treatment includes:

     * Standard doublet chemotherapy
     * Immunotherapy
     * Targeted therapy
     * Palliative radiotherapy
     * Local treatment of oligometastatic disease, including surgery and stereotactic radiotherapy
     * Any combination of the above-mentioned treatment modalities Patients are eligible regardless of whether they at the time of inclusion continue maintenance treatment or not

Exclusion Criteria:

1. Progressive disease at first evaluation scan
2. Persons deprived of liberty or under guardianship or curators
3. Dementia, mental alteration or psychiatric disease that can compromise informed consent from the patient and / or adherence to the protocol and the monitoring of the trial
4. Pregnant or breastfeeding women
5. Patient participating in another interventional study during the surveillance period. This is only relevant for studies that might interfere with the intervention. Participation in protocols related only to treatment will not preclude participation in the present study. Cases of doubt will be settled by the protocol committee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2 years

SECONDARY OUTCOMES:
ECOG (Eastern Cooperative Oncology Group) Performance status at time of progression | 2 years
  (0-5) 0 - Asymptomatic (Fully active, able to carry on all predisease activities without restriction)
  1. - Symptomatic but completely ambulatory (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. For example, light housework, office work)
  2. - Symptomatic, <50% in bed during the day (Ambulatory and capable of all self care but unable to carry out any work activities. Up and about more than 50% of waking hours)
  3. - Symptomatic, >50% in bed, but not bedbound (Capable of only limited self-care, confined to bed or chair 50% or more of waking hours)
  4. - Bedbound (Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair)
  5. - Death
Progression free survival | 2 years
Type of treatment at time of progression | 2 years
  Number of patients who are candidates for 2nd line medical antineoplastic treatment
Quality of life (QOL) measured by EuroQol EQ-5D-5L. | 2 years
  EQ-5D-5L measures individual generic health status using 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, and each dimension has 5 levels depending on severity of symptoms (1 no problems, 5 extreme problems) and a VAS (visual analogue scale). The scores can then be converted into a single index number. The index value will be used for calculation of quality-adjusted life years (QALYs) for a health economic analysis of the intervention.
Quality of life measured by EORTC QLQ C30/LC13. | 2 years
  The EORTC QLQ-C30 questionnaire consists of 30 questions with five functional scores (physical, role, cognitive, emotional and social); a global health status score three symptom scale score (fatigue, pain, nausea and vomiting); and six independent one-item scores describing additional symptoms (dyspnea, appetite loss, sleep disturbance, constipation and diarrhea) and financial burden.
  The EORTC QLQ-LC13 is a supplementary module to the C30 questionnaire and generates a multiple-item scale score of dyspnea and a number of single-item scores that assesses chest pain, arm / shoulder pain, pain in other parts, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia and hemoptysis.
  All scales and single-item scores can be linearly transformed to a score ranged from 0 to 100. A higher score of global health and functional subscriptions indicates better functioning.
HADS score (Hospital Anxiety And Depression Scale) | 2 years
  The HADS (The hospital anxiety and depression scale) is a fourteen-item scale. Seven items relate to depression and seven to anxiety. The tool has been developed for detection of anxiety and depression in patients with physical health problems. All items are scored from 0-3 with a possible total score between 0 and 21 for anxiety and depression respectably.
  A cut-off point of >7 for anxiety or depression is considered significant.
Qualitative interviews | 2 years
  Qualitative interviews with members of the clinical staff and a group of patients in the intervention arm will be conducted during the study period. The purpose is to identify barriers, advantages and possible reasons for the outcomes of the study.
Baseline questionnaires of non-participants | 2 years
  All patients who met the inclusion criteria but declined to participate in the trial will be asked to fill in a questionnaire. The questionnaire will include information on socioeconomics, reasons for non-participation and the same HRQoL questionnaires that are filled in by the participants in the trial (EORTC QLQ-C30/LC13, HADS, EQ-5D-5L).
  The purpose is to identify baseline differences between participants and non-participants and thereby testing the PRO system for generalizability.

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus Friis, MD, Principal Investigator — Department of Oncology, Regional Hospital West Jutland
Locations (1):
- Department of oncology, Regional Hospital West Jutland, Herning, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Friis RB, Pappot H, Hjollund NH, McCulloch T, Holt MI, Persson GF, Wedervang K, Clausen MM, Wahlstrom S, Hansen KH, Rasmussen TR, Dalton SO, Jakobsen E, Linnet H, Skuladottir H; Danish Lung Cancer Group. Remote Symptom Monitoring of Patients With Advanced Lung Cancer (The ProWide Study): A Randomized Controlled Trial. JCO Oncol Pract. 2025 Jun;21(6):813-823. doi: 10.1200/OP-24-00562. Epub 2024 Dec 10. PMID 39657078

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT03608410/Prot_SAP_000.pdf